CLINICAL TRIAL: NCT03744117
Title: Telemedicine Facilitated Palliative Care Consultations in Rural Dialysis Units
Brief Title: Tele-palliative Care in Rural Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Katharine Cheung, Primary Investigator, Assistant Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS 19-0081
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; end-stage kidney disease; supportive care; palliative care; rural health
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): There is a single arm in this study. All patients will be assigned to receive the intervention, which is a palliative care consultation delivered by telemedicine.
  Interventions: Other: Palliative care consultation

INTERVENTIONS:
Other: Palliative care consultation — A palliative care consultation will occur via telemedicine with patients receiving maintenance dialysis.

SUMMARY:
Telemedicine (TM) is an innovative approach that has successfully facilitated palliative care consultations (PCC) in rural settings but not yet in dialysis. In this study, the investigators will deliver telemedicine-facilitated PCC to rural dialysis units leveraging an existing telehealth network.

DETAILED DESCRIPTION:
Training of dialysis personnel: Dialysis staff will meet with the PI to review eligibility, recruitment and consent during a training meeting prior to beginning recruitment. Overview of the study goals and protocol will also be reviewed at quarterly renal dialysis meetings attended by all nephrologists and dialysis nursing supervisors.

Recruitment and informed consent procedures will occur chairside in the dialysis unit and will be performed by study personnel. Participants will complete a single-item Heard and Understood questionnaire and demographic survey with research personnel.

Consented individuals will be contacted by the research team to schedule an appointment via telemedicine. Scheduling of Telemedicine-palliative care consultation (TM-PCC) will occur as per usual care, based on availability of patient and family, clinician and space, and will be coordinated by study personnel with dialysis staff input. Attention will be paid to travel adjustments as necessary for dialysis patients.

PCC will occur at the dialysis unit. The clinician will be located at UVMMC, at a telemedicine station assigned for this task. The palliative care consult can happen during dialysis and using an iPad and headphones may be worn.

The intervention will occur while on dialysis, unless otherwise requested, using an iPad mounted on a portable stand. Dialysis or research staff will open the Zoom application for the patient and the PCC will occur via Zoom, an encrypted service used by UVMMC already for telemedicine. Headsets will be provided to the patient (and family) to cancel out ambient noise and to enhance privacy. Participants can also choose to have the palliative care consult before or after dialysis, or at home, if they have an internet connection.

The consult will be video-recorded in order to analyze the quality of communication and content of palliative care consults in dialysis patients. Most palliative care consults last about one hour. After the consult, participants will complete a questionnaire. This should not take more than 5-10 minutes.

There is only one visit required in this study. If participants desire follow-up with the palliative care team, this can be arranged but is not part of the study. We will assess outcomes at 6 months by reviewing the medical record for any hospitalizations, hospice enrollment, withdrawal from dialysis or other changes to dialysis treatment.

Per usual care, the palliative care clinician will summarize the consult and send this to the nephrologist and/or primary care provider.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 and older, receiving maintenance dialysis who are willing and capable of providing informed consent.

Exclusion Criteria:

* Patients with dementia or other medical conditions that would impair their ability to consent, participate in conversation or complete questionnaires, or patients expected to transfer to a dialysis unit outside of Vermont within 6 months would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Feasibility will be defined as the 1 month completion rate of the consult from time of participant recruitment to the consult. | This will be assessed at 18 months.
  We will define feasibility as the 1 month completion rate of the consult from time of participant recruitment to the consult.
Acceptability :We will measure acceptability of the telemedicine intervention using a 5-point likert scale. | This will be assessed at 18 months.
  We will measure acceptability of the telemedicine intervention using a 5-point likert scale.

SECONDARY OUTCOMES:
Quality of communication reported by patients:Quality of communication will be measured using an adapted form of the Quality of Communication survey tool. This consists of 6 questions, each with a score of 0-10. | The survey will be completed within 2 weeks of the intervention.
  Quality of communication will be measured using an adapted form of the Quality of Communication survey tool. This consists of 6 questions, each with a score of 0-10.
Heard and Understood: Participants will rate on a 5-point scale whether they felt heard and understood during the palliative care consultation. | This question will be completed within 2 weeks of the intervention.
  Participants will rate on a 5-point scale whether they felt heard and understood during the palliative care consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine L Cheung, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung KL, Tamura MK, Stapleton RD, Rabinowitz T, LaMantia MA, Gramling R. Feasibility and Acceptability of Telemedicine-Facilitated Palliative Care Consultations in Rural Dialysis Units. J Palliat Med. 2021 Sep;24(9):1307-1313. doi: 10.1089/jpm.2020.0647. Epub 2021 Jan 19. PMID 33470899

DOCUMENTS (1):
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03744117/ICF_000.pdf